CLINICAL TRIAL: NCT07299045
Title: The Impact of Mindfulness-Based Psychoeducation on Perceived Stress, Intolerance of Uncertainty, and Cognitive Flexibility in Patients With Anxiety Disorders: A Randomized Controlled Trial
Brief Title: The Impact of Mindfulness-Based Psychoeducation on Perceived Stress, Intolerance of Uncertainty, and Cognitive Flexibility in Patients With Anxiety Disorders
Acronym: Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Eda Mert, Principal Investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/369
Record Dates: First submitted 2025-11-23; First posted 2025-12-23 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Anxiety Disorders; Mindfulness; Perceived Stress; Intolerance of Uncertainty; Cognitive Flexibility
Keywords: Anxiety disorders; Mindfulness; Perceived Stress; Intolerance of Uncertainty; Cognitive Flexibility
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Masking Description: Since the intervention component of the study included tangible elements such as training and counseling, it was not possible to blind participants or researchers to group allocation. The assignment of participants to groups was carried out by the researchers without blinding. Data for the personal information form and all dependent variables of the study were collected through self-report at both the pretest and posttest stages, and in this respect, the researchers were blinded to the scale results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants receive a structured mindfulness-based psychoeducation programin addition to standard care. The intervention includes psychoeducational sessions, mindfulness exercises, and practical strategies.
  Interventions: Other: Mindfulness-Based Psychoeducational Program
- Control (No Intervention): Participants receive standard care only without any additional psychoeducational or mindfulness-based intervention.

INTERVENTIONS:
Other: Mindfulness-Based Psychoeducational Program — Mindfulness-Based Psychoeducational Program contains 8-sessions named as "Introduction to mindfulness, Exploring Mindfulness, Becoming Mindful of the Autopilot, Being in the Body, Meeting Stress with Mindfulness, Mindful Communication, Staying with Difficulties, A New Beginning"
  Arms: Intervention

SUMMARY:
Mindfulness-based interventions, which cultivate the capacity to remain present with difficult thoughts and emotions and to maintain psychological well-being in the face of such challenges, have been shown to facilitate positive change in individuals with anxiety disorders. The present study aimed to investigate the effects of a mindfulness-based psychoeducational program on perceived stress, intolerance of uncertainty, and cognitive flexibility among individuals diagnosed with anxiety disorders.

This randomized controlled trial with pre-test, post-test, and one-month follow-up measurements was conducted with individuals who applied to the Psychiatry Outpatient Clinic at Aydın Atatürk State Hospital and were diagnosed with anxiety disorders. A total of 50 participants were included in the study and were randomly assigned to groups (Experimental: 25; Control: 25). The experimental group underwent an 8-week mindfulness-based psychoeducational program, while no intervention was provided to the control group. Research data were collected using the Personal Information Form, Perceived Stress Scale (PSS), Intolerance of Uncertainty Scale (IUS-12), and Cognitive Flexibility Scale (CFS).

ELIGIBILITY:
Inclusion Criteria:

* Being literate
* Having a diagnosed anxiety disorder
* Being 18 years of age or older

Exclusion Criteria:

* Presence of an acute episode of the illness
* Lack of ability to engage in communication
* currently receiving another form of psychotherapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | Pre-test; post-test (at the end of 8-week psychoeducational program); 1-month follow-up test
  Differences in participants' perceived stress levels pre- and post-psychoeducation. Higher scores obtained from the scale indicate greater levels of perceived stress.
Intolerance of Uncertainty Scale | Pre-test; post-test (at the end of 8-week psychoeducational program); 1-month follow-up test
  Differences in participants' intolerance of uncertainty levels pre- and post-psychoeducation. Higher scores obtained from the scale indicate greater levels of intolerance of uncertainty.
Cognitive Flexibility Scale | Pre-test; post-test (at the end of 8-week psychoeducational program); 1-month follow-up test
  Differences in participants' cognitive flexibility levels pre- and post-psychoeducation. Higher scores on the scale indicate higher levels of cognitive flexibility.

CONTACTS AND LOCATIONS:
Locations (1):
- Eda Mert, Aydin, Turkey (Türkiye)